CLINICAL TRIAL: NCT05938400
Title: Clinical Evaluation of Impressions Made Using One Step & Two Step Polyvinylsiloxane Impression Techniques and Resulting Fixed Prosthesis-A Randomised Controlled Trial
Brief Title: Impression & Prosthesis Quality Made From Different Polyvinylsiloxane Impression Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Humera Nasim, Lecturer (Prosthodontics department), Principal investigator, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2932
Record Dates: First submitted 2023-03-25; First posted 2023-07-10 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Endodontically Treated Teeth; Missing Teeth; Discoloration, Tooth; Prosthesis Failure, Dental; Open Margin on Tooth Restoration
Keywords: Polyvinylsiloxane impression; fixed prosthetics; impression techniques; single stage impression; two step putty wash impression; marginal fit; prosthesis fit; endodontically treated teeth
MeSH Terms: conditions — Tooth, Nonvital; Anodontia; Tooth Discoloration; Prosthesis Failure

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- One step polyvinylsiloxane impression technique (Experimental): All impressions in this group will be recorded in a single stage, mixing light-bodied PVS material and putty PVS material simultaneously and recording of impression of prepared tooth
  Interventions: Device: Polyvinylsiloxane impression with different techniques
- Two step polyvinylsiloxane impression technique (Active Comparator): All impressions in this group will be made in two stages, recording putty PVS impression first and then reloading it with light-bodied PVS material to record final impression.
  Interventions: Device: Polyvinylsiloxane impression with different techniques

INTERVENTIONS:
Device: Polyvinylsiloxane impression with different techniques — One step impression technique will be compared with the standard two step technique

SUMMARY:
This randomized controlled trial is to clinically assess and compare impression quality of polyvinylsiloxane impression material using one step (experimental) and two step (control) impression techniques and its effect on marginal fit of prosthesis and proximal contact of prosthesis.

DETAILED DESCRIPTION:
Study participants will be randomly allocated to either of the two groups (experimental or control) through software-generated random numbers.

Indicated tooth will be prepared to receive a fixed prosthesis under local anesthesia as per standard guidelines.

Polyvinylsiloxane (PVS) impressions will be recorded in stock tray after moisture control, according to the assigned group.

In experimental group, light body and putty PVS will be mixed simultaneously and placed in stock tray to record impressions in single stage.

In control group, a putty PVS impression will be recorded first in stock tray and allowed to set. After setting of putty PVS, light-bodied PVS material will be applied to recorded impression surface and reseated in mouth to record final impression in second stage.

All impressions will be disinfected according to the recommended guidelines. All impressions will then be assessed by a senior clinician using 3.5 x magnification loupe and graded according to the selected criteria.

Impressions will then be poured in dental stone and prosthesis will be manufactured in dental lab.

Participants will be recalled for prosthesis trial and fit assessment of prosthesis margins using a dental explorer instrument and visual evaluation. Proximal contact of prosthesis will be graded according the criteria and assessed using dental floss.

Satisfactory prostheses will be cemented after final adjustments.

ELIGIBILITY:
Inclusion Criteria:

* Indication of fixed-fixed partial denture or crown
* Good oral hygiene
* Sound abutment tooth (vital/non-vital)

Exclusion Criteria:

* Failure to provide written consent to participation in study
* Long span bridges (Greater than 3 units)
* Patients with bleeding disorders
* Cases indicated for resin-bonded prosthesis

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2023-07-02 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Incidence of defects in impression recorded to fabricate dental prosthesis as assessed by impression quality assessment scale | 10 minutes
  Outcome assessment scale: 1. Perfect impression, no voids or defects; 2. Acceptable impression, minimal defects in non critical region; 3. Unacceptable impression, defects involving critical region.

SECONDARY OUTCOMES:
Incidence of prosthesis margin defects as assessed by Marginal adaptation assessment scale | 14 days
  Outcome assessment scale: 1. Adequate, adapted to tooth margins; 2. Inadequate, not accurately adapted to tooth margin
Incidence of prosthesis proximal contact inaccuracy as assessed by prosthesis contact assessment scale | 14 days
  Outcome assessment scale: 1. Acceptable, same as natural proximal contact on contralateral side; 2. Unacceptable; either tight or open proximal contact.

CONTACTS AND LOCATIONS:
Locations (1):
- Dow University of Health Sciences, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No